CLINICAL TRIAL: NCT04584164
Title: Interest of the Sialendoscopy Associated With a Local Injection of Corticosteroids in the Treatment of Radio-induced Xerostomia in Comparison With the Hygiene Rules: a Prospective Randomized and Controlled Study
Brief Title: Interest of the Sialendoscopy Associated With a Local Injection of Corticosteroids in the Treatment of Radio-induced Xerostomia in Comparison With the Hygiene Rules
Acronym: SIALORAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIALORAD
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Xerostomia
Keywords: xerostomia; sialendoscopy; corticosteroids; ENT
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: The study aims at comparing the sialendoscopy associated with a local injection of corticosteroids to the basic hygiene rules in the treatment of Xerostomia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): This arm involves patients applying the basic hygiene rules (with mouthwashes) without the sialendoscopy method.
- Sialendoscopy arm (Experimental): This arm involves patients applying the hygiene rule and benifiting in addition a sialendoscopy treatment with a local injection of corticostéroïdes (at the end of the procedure) in the treatment for Xerostomia.
  Interventions: Device: sialendoscopy

INTERVENTIONS:
Device: sialendoscopy — The patients applying the hygiene rule and benifiting in addition a sialendoscopy treatment with a local injection of corticostéroïdes (at the end of the procedure) in the treatment for Xerostomia.
  Arms: Sialendoscopy arm

SUMMARY:
Xerostomia is defined as the subjective sensation of dry mouth, and may be associated with a reduction in saliva secretion and composition. It is one of the most common complaints found in patients after irradiation in the head and neck area. This complaint is found in a large majority of patients during radiotherapy, continuing for several years after stopping radiotherapy (93% during radiotherapy and 40 to 60% after two years post-radiotherapy). The advent of IMRT (Intensity-Modulated Radiation Therapy) has reduced this complaint, but it still concerns 40% of patients undergoing post-radiotherapy affecting the head and neck. Xerostomia is responsible for pronunciation difficulties, dysphagia, dysgeusia, alteration of the oral condition leading to a significant alteration of the quality of life. This complaint is maximal in the first six months following radiotherapy, then stabilizes or even regresses in the year following radiotherapy but can persist well beyond the end of the irradiation. At present, there are few treatments that have been shown to be truly effective. Systemic treatments (sialogues, cholinergic agonists, parasympathomimetic and muscarinic agonists, corticosteroids, etc.) allow partial improvement with delayed and not prolonged effectiveness. Many studies evaluating the efficacy of these therapies have shown contradictory and insufficient results (less than half of the patients present an improvement under treatment), without ever allowing a complete cure. Surgical treatments by submaxillary gland transfer have also been studied, but at the price of significant morbidity (cervicotomy, risk to the chin nerve in post-radial areas, etc.). Conformational radiotherapy with intensity modulation has made it possible to reduce the severity of xerostomia but does not make it possible to free oneself from this complication. Patients often find themselves reduced to symptomatic adjunctive treatments (gland massage, sprays, hydration, acupuncture...) without curative treatment. There is therefore a real need to respond to the complaint expressed by many patients by proposing an effective and long-lasting therapy.

DETAILED DESCRIPTION:
Post-radiation xerostomia appears from the first days after irradiation and for very low doses (from a dose received of 5 Gy). A first phase appears in the first 10 days following radiotherapy, with regression of salivary secretion by blocking the muscarinic membrane receptors of acinar cells and destruction of the endothelial cells responsible for glandular angiogenesis. With increasing doses, apoptosis of stem cells and acinar cells of the salivary glands follows, leading to atrophy and irreversible fibrosis beyond 60 Gy, due to the lack of renewal of acinar stem cells. Four phases in the pathophysiology of post-radial xerostomia are thus described. Phases 1 and 2, appearing respectively between 0-10 days and 10-60 days, are characterized by a severe decrease in saliva production, first without a decrease in amylase production or in the number of acinar cells in phase 1 and then with a decrease in amylase and in the number of acinar cells in phase 2. This acute phase, initially reversible, is thought to be related either to apoptosis of acinar cells or to acinar cell membrane dysfunction. Then phases 3 and 4, appearing respectively between 60-120 days (stability of the secretion and number of acinar cells) and between 120 and 240 days, are characterized by a senescence of mature acinar cells, which are not renewed due to sterilization of the glandular stem cells, leading to a definitive deterioration of the secretory functions by glandular atrophy and irreversible fibrosis. A study by the QUANTEC (Quantitative Analyses of Normal Tissue Effects in the Clinic) group showed that severe xerostomia (defined as a decrease of more than 25% in the amount of saliva produced) could be seen in IMRT when the four major salivary glands were given a dose >25Gy or if at least one parotid gland was not preserved at a dose <20Gy. The pathophysiology of post-radial xerostomia has similarities with that of other causes of xerostomia. Gougerot-Sjögren's syndrome is characterized by salivary gland infiltration by B and T macrophages and lymphocytes targeting salivary muscarinic receptors. This is followed by inflammation and lymphocytic infiltration with replacement of glandular acinar cells by fibrosis associated with cellular apoptosis and thus glandular atrophy. The complaint of xerostomia and objective reduction of saliva secretion are frequently found in post-irradiation therapy, used for the treatment of thyroid cancer. Indeed, salivary glandular cells have a strong affinity for Iodine-131 leading to inflammation of the ductal epithelium and endothelial cells, resulting in ductal and glandular fibrosis. These pathophysiological changes during Gougerot-Sjögren and post-irradiotherapy are correlated with sialendoscopic findings: stenosis, sialadenitis, sialadochitis, mucous plugs, erythema... . However, studies have shown the effectiveness of sialendoscopy in improving the symptomatology of xerostomia and in increasing salivary production, by simple irrigation (of serum alone or associated with local injection of corticosteroids) and root canal dilatation in patients with these non-lithiasic pathologies. Therapeutic success would be attributable to the removal of mucosal plugs, removal of stenosis and reduction of inflammation (25). This is all the more so since the saliva flow produced by the acinar cells and the salivary ionic composition (by ductal ionic reabsorption) are strongly dependent on the ductal flow, and therefore on the presence of possible stenosis or mucous plugs. The improvement of the symptomatology and salivary production would be visible in the immediate postoperative period (from the first weeks), with a prolonged therapeutic effect beyond several months, after a single sialendoscopy. Recently, a study has shown the efficacy of sialendoscopy to improve chemotherapy-induced xerostomy symptoms using Ac-PSMA-617 for the treatment of prostate cancer, which is also the cause of Grade 1 xerostomia. Our study is based on the pathophysiological similarity of post-radial xerostomy with Gougerot-Sögren's syndrome and post-irradial xerostomy. The promising results of recently published sialendoscopic studies in these two pathologies allow us to envisage a potential benefit of sialendoscopy in a post-radial context.

In the context of this work, the investigators will compare sialendoscopy associated with a local injection of corticosteroids to the usual management based on the hygieno-dietary rules (HDR) consisting of regular drinking and a diet with a high dose of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years old
* Negative pregnancy test for women of childbearing age
* Patient with head and neck cancer who has had parotid and submaxillary gland irradiation at a received dose greater than or equal to 60 Gy and whose end of treatment by radiotherapy is less than 6 months.
* Patient with a complaint of xerostomia/dry mouth ≥1 month and wishing to benefit from therapeutic treatment
* Patient affiliated to a social security system
* Francophone patient
* Patient who has given free, informed and written consent.

Exclusion Criteria:

* History of surgery of the 4 salivary glands (parotidectomy, under maxillectomy, pelvectomy) or prior sialendoscopy
* Current episode of submaxillitis or acute infectious parotitis
* Presence of a lithiasis pathology on the post-radiotherapy control CT scan
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Pregnant or nursing patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Superiority of sialendoscopy combined with local injection of corticosteroids (intervention group) in improving the symptoms of post-radial xerostomia, compared to the usual HDR-based treatment | 6 months
  Difference in mean scores of the Xerostomia Questionnaire (XQ) 6 months after the start of treatment between the 2 groups of patients.

SECONDARY OUTCOMES:
To compare the efficacy of sialendoscopy associated with local corticosteroid injection compared to the usual HDR-based treatment on the early improvement of patient-reported symptoms of post-radial xerostomia | 1 month
  Difference between the two groups of patients in the mean of the Xerostomia Self Questionnaire scores 1 month after the start of treatment
To compare the efficacy of sialendoscopy associated with a local corticosteroid injection compared to usual HDR-based treatment on the prolonged improvement of post-radial xerostomy symptoms reported by patients. | 1 year
  Difference between the two groups of patients in the mean scores of the Xerostomia Questionnaire (XQ)1 year after the start of treatment
To compare the effectiveness of sialendoscopy associated with a local corticosteroid injection compared to that of standard HHR-based treatment in improving quality of life. | 1 month
  Difference between the two groups of patients in the mean of the Quality of Life Self Questionnaire (EORTC-QLQ-C30 HN35) scores 1 month after the start of treatment
To compare the effectiveness of sialendoscopy associated with a local corticosteroid injection compared to the usual HDR-based treatment on the improvement of stimulated and non-stimulated saliva production. | 1 month
  Difference between the two groups of patients in the mean amount of saliva produced stimulated and unstimulated (sialometry) 1 month after the start of treatment
To compare the efficacy of sialendoscopy associated with local corticosteroid injection compared to usual HDR-based treatment on the improvement of post-radial xerostomy symptoms reported by patients according to the rate of salivary gland irradiation. | 1 month
  Difference between the two groups of patients in the mean of the Xerostomia Self-Dose Questionnaire scores by site in Gy (dose-volume histograms) 1 month after the start of treatment.
To compare the efficacy of the intervention group compared to the usual HDR-based treatment on the improvement of stimulated and non-stimulated saliva production according to the rate of irradiation of the salivary glands. | 1 month
  Difference between the two groups of patients in the average amount of saliva produced stimulated and unstimulated (sialometry) as a function of the dose received in Gy (dose-volume histograms) 1 month after the start of treatment
Describe the post-radial sialendocopic appearance at the parotid and submaxillary levels. | Day 1
  In patients in the sialendoscopy group: intraoperative aspects of the extra and intraglandular parotid and submaxillary salivary ducts in sialendoscopy: stenosis, lithiasis, mucous plug, inflammation, erythema, pallor.
Describe post sialendoscopy complications in this field | 1 month
  In patients in the sialendoscopy group: frequency of complications of sialendoscopy. Complications are classified as minor (pain, oedema, infection, hemorrhage, paresthesia of the lingual nerve) or major (need to return to the operating room, death), with their duration of early (if ≤ 7 days postoperatively) or delayed (≤ 30 days) onset.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth SAUVAGET, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France